CLINICAL TRIAL: NCT07359989
Title: Leucine Combined With Radiotherapy and Chemotherapy as Neoadjuvant Therapy for Locally Advanced Rectal Cancer: A Single-Arm Clinical Study
Brief Title: Leucine Plus Radiochemotherapy for Neoadjuvant Treatment of Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Qichun Wei, MD, PhD, Second Affiliated Hospital, School of Medicine, Zhejiang University, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT 2025-0428
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-03

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Leucine
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leucine plus Radiotherapy and Chemotherapy (Experimental): Leucine plus radiotherapy and chemotherapy as neoadjuvant therapy
  Interventions: Dietary Supplement: Oral administration of Leucine

INTERVENTIONS:
Dietary Supplement: Oral administration of Leucine — Oral administration of leucine during radiotherapy

SUMMARY:
Colorectal cancer (CRC), a prevalent gastrointestinal malignancy, is experiencing a rising incidence in China. Rectal cancer constitutes nearly half of all new CRC cases, with over half of these patients diagnosed at a locally advanced stage. While neoadjuvant chemoradiotherapy is the standard of care for these patients, it yields a pathological complete response in only 10-30% of cases, and the risk of recurrence and metastasis remains suboptimal.

The role of amino acid metabolism in cancer therapy is gaining significant interest. Our preliminary data reveal that leucine-derived metabolite significantly impairs cellular DNA damage repair and enhances the efficacy of radiotherapy. However, it remains unknown whether combining leucine with chemoradiotherapy can improve tumor regression and survival in patients with locally advanced rectal cancer.

The goal of this single-arm clinical trial is to evaluate the safety and efficacy of Leucine combined with neoadjuvant chemoradiotherapy for locally advanced rectal cancer, potentially offering a new therapeutic option.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily participates in this study, signs the Informed Consent Form, demonstrates good compliance, and cooperate with follow-up;
2. Aged 18 to 80 years (inclusive), both male and female are eligible;
3. Histologically confirmed and assessed as locally advanced rectal adenocarcinoma (confirmed by MRI): cT3 or higher; or cN+;
4. MRI confirms that the lower edge of the tumor is ≤10 cm from the anal verge;
5. No prior anti-tumor treatment for rectal cancer (except for traditional Chinese medicine treatments);
6. ECOG score of 0-1;
7. Major organs or functions meet the following criteria (within 2 weeks before the test, no use of any blood components or growth factors for correction is allowed):

   Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelets ≥100×10^9/L; Hemoglobin ≥10 g/dL; Serum albumin ≥3.0 g/dL; Total bilirubin ≤ ULN, ALT, AST, and/or AKP ≤2.5 × ULN; Serum creatinine ≤ ULN or creatinine clearance rate ≥60 mL/min; International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ ULN;
8. Female patients of childbearing potential must agree to abstain from heterosexual intercourse or use reliable and effective contraception from the time of signing the informed consent form until at least 6 months after the last dose of study drug. A serum HCG test must be negative within 7 days before starting treatment, and the woman must not be breastfeeding. A woman is considered of childbearing potential if she has had menstruation, has not reached postmenopausal status (absence of menstruation for ≥12 consecutive months without any other cause), and has not undergone sterilization surgery (such as hysterectomy, bilateral tubal ligation, or bilateral oophorectomy);
9. Male patients with female partners of childbearing potential must agree to abstain from intercourse or use reliable and effective contraception from the time of signing the informed consent form until at least 6 months after the last dose of study drug. Male patients must also agree not to donate sperm during this period. Male patients with pregnant partners should use a condom, without the need for additional contraceptive methods.

Exclusion Criteria:

1. Patients with locally recurrent rectal cancer after previous treatment;
2. Patients assessed by the investigator as having initially unresectable rectal cancer or those deemed unable to tolerate surgery;
3. Clinical or imaging evidence suggests distant metastasis or positive lateral lymph nodes;
4. Patients with multiple colorectal cancer lesions;
5. Clinical or imaging evidence suggests bowel obstruction or perforation, or the investigator evaluates a high risk of perforation or bleeding;
6. Factors deemed by the investigator to make the patient unsuitable for long-course radiotherapy;
7. Severe cardiovascular or cerebrovascular diseases, including cerebrovascular accident (CVA), transient ischemic attack (TIA), myocardial infarction, or significant vascular disease (such as an aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to enrollment; poorly controlled cardiac symptoms or diseases, such as unstable angina, NYHA class II or higher heart failure, left ventricular ejection fraction <50% by echocardiography, or severe arrhythmias not controlled by medication;
8. History of active pulmonary tuberculosis detected by medical history or CT, active pulmonary tuberculosis within 1 year before enrollment, or a history of active tuberculosis more than 1 year ago that was not properly treated;
9. Major surgery within 3 months before starting study treatment (major surgery is defined as surgery performed under general anesthesia); presence of non-healing wounds (severe, non-healing or dehiscent), active peptic ulcers, or untreated fractures;
10. Difficulty swallowing or other factors affecting oral medication use;
11. Contraindications to MRI;
12. Active autoimmune disease or history of autoimmune diseases (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, colitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [patients controlled by thyroid hormone replacement therapy can be included]); patients with skin diseases that do not require systemic treatment (e.g., vitiligo, psoriasis, alopecia), controlled type 1 diabetes treated with insulin, and childhood asthma that has fully resolved and requires no intervention in adulthood may be included (patients requiring bronchial dilation for asthma cannot be included);
13. History of immunodeficiency, including positive HIV test, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation or allogeneic bone marrow transplantation;
14. Severe infections within 4 weeks before the first use of the study drug (CTCAE > Grade 2), such as severe pneumonia, bacteremia, or infections requiring hospitalization; active lung inflammation on baseline chest imaging, signs and symptoms of infection requiring oral or intravenous antibiotics within 2 weeks before the first use of the study drug, except for prophylactic antibiotics;
15. Current or past history of interstitial lung disease or interstitial pneumonitis requiring steroid therapy, or other conditions (e.g., lung fibrosis, organizing pneumonia such as bronchiolitis obliterans) that may interfere with the assessment and management of immune-related lung toxicity, evidence of active pneumonia on screening chest CT, or severely impaired lung function;
16. Active hepatitis B (HbsAg positive, and HBV-DNA ≥ 2,500 copies/ml or 500 IU/ml) or active hepatitis C (HCV antibody positive and HCV-RNA above the detection limit); co-infection with hepatitis B and hepatitis C (HbsAg or HbcAb positive and HCV antibody positive);
17. Diagnosis of another malignancy within 5 years prior to the first use of the study drug (patients with effectively treated basal cell carcinoma, squamous cell carcinoma of the skin, and/or effectively excised in situ cervical or breast cancer may be included upon evaluation, but those who previously received immunotherapy, chemotherapy, targeted therapy, or radiation therapy cannot be included);
18. Known allergy, hypersensitivity, or contraindications to pucotenlimab, oxaliplatin, capecitabine, or any component of their formulations;
19. Use of immunosuppressants or corticosteroids (dose >10 mg/day prednisone or equivalent) for immunosuppression within 14 days before starting study treatment; inhaled or topical steroids are allowed in the absence of active autoimmune disease, and hormone replacement therapy with ≤10 mg/day prednisone or equivalent is permitted;
20. Participation in another clinical study within 4 weeks before the first use of the study drug (for participants in the follow-up phase of another study, the time is calculated from the last use of investigational drug or device);
21. Laboratory abnormalities of sodium, potassium, or calcium greater than Grade 1 within 2 weeks before the start of study treatment that cannot be corrected with treatment;
22. Receipt of live attenuated vaccines within 28 days before starting study treatment or planning to receive such vaccines during the treatment period or within 60 days after the last dose of the study drug;
23. Pregnant or breastfeeding women;
24. Any other factors, as judged by the investigator, that may affect the study results or lead to premature termination, such as alcohol abuse, drug abuse, other serious diseases (including mental disorders) requiring concomitant treatment, severe laboratory abnormalities, family or social factors, and other conditions that may affect participant safety or data collection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The Pathological complete response (pCR) rate | From enrollment to the end of treatment at 16 weeks.
  The definition of pCR is that after surgery, in the pathological evaluation of the resected rectal cancer lesion, mesorectum, and regional lymph node samples, there are no visible tumor cells under the microscope. Tumor cells refer to viable tumor cells, excluding degenerated or necrotic cells. Pools of acellular mucin should not be assessed as residual tumor.
Clinical complete response (cCR) rate | From enrollment to the end of treatment at 12 weeks.
  The cCR assessment is defined by the fulfillment of the following three criteria:
  1. Digital rectal examination of the original tumor area shows normal findings, with no palpable tumor masses.
  2. Endoscopy reveals white, flat mucosal scars accompanied by surrounding capillary ectasia, without evidence of tumor ulcers or nodules; mucosal biopsy results are negative for cancer cells.
  3. Contrast-enhanced MRI of the rectum shows: On T2-weighted images, only low signal intensity (dark on T2) is present without intermediate T2 signal intensity, and there are no signs of enlarged lymph nodes. there is no visible signal on diffusion-weighted (DW) images.

SECONDARY OUTCOMES:
Adverse events. | From enrollment to the end of treatment at 3 years.
  The incidence, type, and severity of adverse events (AEs), serious AEs, and immune-related AEs (irAEs) were assessed in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE version 5.0).
The rate of TRG0 | From enrollment to the end of treatment at 16 weeks
  Complete regression, defined as no residual tumor cells in the primary tumor and regional LNs (ypT0N0)
The rate of R0 resection | From enrollment to the end of treatment at 16 weeks.
  R0 resection is defined as the removal of the rectal cancer lesion during surgery with no tumor cells present within 1 mm of the resection margins.
Event-Free Survival | From enrollment to the end of treatment at 3 years
  Event-Free Survival (EFS) was defined as the period from the date of first treatment administration to the date of the first documented relevant event, where relevant events include disease progression that leads to inoperability, local recurrence or distant metastasis after surgery, and death due to any cause.
Overall Survival | From enrollment to the end of treatment at 3 years
  OS (Overall Survival) is defined as the period from the date of first treatment administration to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital Of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No